CLINICAL TRIAL: NCT05624710
Title: A Phase 1, Open-Label Study to Evaluate the Pharmacokinetics and Safety of INCB054707 in Participants With Normal Hepatic Function and Participants With Hepatic Impairment
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of INCB054707 in Participants With Normal Hepatic Function and Participants With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 54707-105; 2022-002660-70 (EudraCT Number)
Record Dates: First submitted 2022-11-11; First posted 2022-11-22 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Renal Insufficiency; Kidney Diseases
Keywords: renal impairment; hemodialysis; Kidney failure; end-stage renal disease
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases; Kidney Failure, Chronic

STUDY DESIGN:
Masking Description: open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: Severe Hepatic Impairment (Experimental): Participants with severe hepatic impairment (Class C Child-Pugh score) will receive a single oral dose of INCB054707 on Day 1.
  Interventions: Drug: INCB054707
- Group 2: Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment (Class B Child-Pugh score) will receive a single oral dose of INCB054707 on Day 1.
  Interventions: Drug: INCB054707
- Group 3: Mild Hepatic Impairment (Experimental): Participants with mild hepatic impairment (Class A Child-Pugh score) will receive a single oral dose of INCB054707 on Day 1.
  Interventions: Drug: INCB054707
- Group D: Normal Hepatic Function (Experimental): Participants with normal hepatic function will receive a single oral dose of INCB054707 on Day 1.
  Interventions: Drug: INCB054707

INTERVENTIONS:
Drug: INCB054707 — INCB054707 75 mg will be administered orally on Day 1.
  Other Names: Povorcitinib

SUMMARY:
This is a multicenter, open-label, parallel-group study to evaluate INCB054707 in participants with varying levels of renal function or impairment.

ELIGIBILITY:
Inclusion Criteria:

- Participants with hepatic impairment will be classified at screening based on Child-Pugh score. Classification will be repeated at check-in and should not be significantly different.

If the hepatic function classification for the participant is not similar at the 2 timepoints, enrollment of the participant into a hepatic category group will be at the discretion of the investigator, in consultation with the sponsor's medical monitor. The enrollment group will be based on the results at screening.

* Participants eligible for Group 4 (normal hepatic function) should be in good health as determined by no clinically significant findings in the medical history, physical examination, vital signs, 12-lead ECGs, or laboratory examinations at screening or check-in.
* Participants eligible for Groups 1 through 3 may have medical findings consistent with their degree of hepatic dysfunction, as determined by medical history, physical examination, vital signs, 12-lead ECGs, and clinical laboratory examinations at screening and check-in. Participants with abnormal findings considered not clinically significant by the investigator are eligible.
* BMI within the range of 18.0 to 44.0 kg/m2 (inclusive) at screening.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* the opinion of the principal investigator, history of uncontrolled or unstable cardiovascular, respiratory, renal, GI, endocrine, hematopoietic, psychiatric, and/or neurological disease within 6 months of screening or evidence of rapidly deteriorating hepatic function.
* Serum corrected calcium and phosphorus levels over the upper limits of the institutional normal ranges.
* History or current diagnosis of uncontrolled or significant cardiac disease indicating significant risk of safety for participation in the study, including any of the following:

  1. Recent myocardial infarction (within 6 months of check-in).
  2. New York Heart Association Class III or IV congestive heart failure.
  3. Unstable angina (within 6 months of check-in).
  4. Clinically significant (symptomatic) cardiac arrhythmias (eg, sustained ventricular tachycardia, second or third degree atrioventricular block without a pacemaker).
  5. Uncontrolled hypertension.
* A current, functioning organ transplant or a scheduled organ transplant in the next 6 weeks from check-in.
* History of malignancy within 5 years of screening, with the exception of cured basal cell carcinoma, squamous cell carcinoma of the skin, ductal carcinoma in situ, or Gleason 6 prostate cancer.
* History of clinically significant GI disease or surgery (cholecystectomy and appendectomy are allowed) that could impact the absorption of study drug.
* Severe ascites (ascites requiring paracentesis more than every 4 weeks) or an encephalopathy ≥ Grade 2 (precludes them from understanding and signing an informed consent).
* Any major surgery within 4 weeks of screening.
* Donation of blood to a blood bank within 4 weeks of screening (within 2 weeks for plasma only).
* Blood transfusion within 4 weeks of check-in.
* Current or recent history (within 30 days before screening) of a clinically significant bacterial, fungal, parasitic, or mycobacterial infection, or currently receiving systemic antibiotics or current clinically significant viral infection at screening or check-in.
* Positive serology for HBV (eg, HBsAg) or HIV. Participants whose results are compatible with immunity due to infection or prior immunization for HBV may be included at the discretion of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Parameter: Cmax of INCBC054707 | Days 1 - 5
  Defined as maximum observed plasma concentration of INCB054707
Pharmacokinetics Parameter: AUC(0-t) of INCB054707 | Days 1 - 5
  Defined as the area under the concentration- time curve up to the last measurable concentration of INCB54707.
Pharmacokinetics Parameter: AUC(0-∞) of INCB054707 | Days 1 - 5
  Defined as area under the concentration-time curve From 0 to Infinity of INCB054707

SECONDARY OUTCOMES:
Number of Treatment Emergent Adverse Events (TEAE'S) | up to 15 days
  Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment.
Pharmacokinetics Parameter: tmax of INCB054707 | Days 1 - 5
  Defined as time to reach maximum plasma concentration of INCB054707
Pharmacokinetics Parameter: t1/2 0f INCB054707 | Days 1 - 5
  Defined as apparent terminal phase disposition half-life of INCB54707
Pharmacokinetics Parameter: CL/F of INCB054707 | Days 1 - 5
  Defined as oral dose clearance of INCB054707
Pharmacokinetics Parameter:: Vz/F of INCB054707 | Days 1 - 5
  Defined as apparent oral dose volume of distribution of INCB054707

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Orange County Research Center, Tustin, California
  - Orlando Clinical Research Center, Orlando, Florida
  - Texas Liver Institute Tli the Liver Institute of South Texas List Downtown Office, San Antonio, Texas
- Apex Gmbh, Munich, Germany

IPD SHARING:
Plan to Share IPD: No